CLINICAL TRIAL: NCT03808493
Title: A Randomized, Open-Label, Single-Dose, 2×2 Crossover Phase 1 Study to Evaluate the Bioequivalence of TAK-438 OD (Orally Disintegrating) 20 mg Tablet When Administered Without Water (Study 1) or With Water (Study 2) and TAK-438 20 mg Tablet When Administered With Water in Japanese Healthy Volunteer Male Subjects
Brief Title: A Bioequivalence (BE) Study of TAK-438 Orally Disintegrating (OD) Tablet
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: TAK-438ODT-1001; U1111-1225-5005 (Other: WHO); JapicCTI-194587 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2019-01-16; First posted 2019-01-17 (Actual); Results first posted 2020-03-24 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-03

CONDITIONS: Japanese Healthy Adult Male
Keywords: Drug Therapy
MeSH Terms: interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Study 1, TAK-438 OD + TAK-438 (Experimental): One TAK-438 OD 20 mg tablet, orally without water under fasted condition, on Period 1 Day 1 in Study 1 (Day 1), followed by a wash-out period (Days 2 to 8), followed by one TAK-438 20 mg tablet, orally with water under fasted condition, on Period 2 Day 1 in Study 1 (Day 9).
  Interventions: Drug: TAK-438 OD; Drug: TAK-438
- Study 1, TAK-438 + TAK-438 OD (Experimental): One TAK-438 20 mg tablet, orally with water under fasted condition, on Period 1 Day 1 in Study 1 (Day 1), followed by a wash-out period (Days 2 to 8), followed by one TAK-438 OD 20 mg tablet, orally without water under fasted condition, on Period 2 Day 1 in Study 1 (Day 9).
  Interventions: Drug: TAK-438 OD; Drug: TAK-438
- Study 2, TAK-438 OD + TAK-438 (Experimental): One TAK-438 OD 20 mg tablet, orally with water under fasted condition, on Period 1 Day 1 in Study 2 (Day 1), followed by a wash-out period (Days 2 to 8), followed by one TAK-438 20 mg tablet, orally with water under fasted condition, on Period 2 Day 1 in Study 2 (Day 9).
  Interventions: Drug: TAK-438 OD; Drug: TAK-438
- Study 2, TAK-438 + TAK-438 OD (Experimental): One TAK-438 20 mg tablet, orally with water under fasted condition, on Period 1 Day 1 in Study 2 (Day 1), followed by a wash-out period (Days 2 to 8), followed by one TAK-438 OD 20 mg tablet, orally with water under fasted condition, on Period 2 Day 1 in Study 2 (Day 9).
  Interventions: Drug: TAK-438 OD; Drug: TAK-438

INTERVENTIONS:
Drug: TAK-438 OD — TAK-438 OD tablet
Drug: TAK-438 — TAK-438 tablet

SUMMARY:
The purpose of this study is to evaluate the BE of single oral dose of TAK-438 OD 20 milligram (mg) tablet without water and TAK-438 20 mg tablet with water (Study 1), and TAK-438 OD 20 mg tablet with water and TAK-438 20 mg tablet with water (Study 2) in Japanese healthy adult male participants.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-438 OD tablet. TAK-438 OD tablet is being tested in Japanese healthy adult men. This study will evaluate bioequivalence of single oral dose of TAK-438 OD 20 mg tablet without water and TAK-438 20 mg tablet with water (Study 1), and TAK-438 OD 20 mg tablet with water and TAK-438 20 mg tablet with water (Study 2).

The study will enroll up to 144 participants in total (Study 1 + 2). In Study 1 and 2, participants will be randomly assigned (by chance, like flipping a coin) to one of the two treatment groups;

Study 1:

* TAK-438 OD 20 mg tablet without water (Period 1) + TAK-438 20 mg tablet with water (Period 2)
* TAK-438 20 mg tablet with water (Period 1) + TAK-438 OD 20 mg tablet without water (Period 2)

Study 2:

* TAK-438 OD 20 mg tablet with water (Period 1) + TAK-438 20 mg tablet with water (Period 2)
* TAK-438 20 mg tablet with water (Period 1) + TAK-438 OD 20 mg tablet with water (Period 2)

This single-center trial will be conducted in Japan. The overall time to participate in this study is approximately 11 days. Participants will make two visits to the clinic and be hospitalized for four days each in Periods 1 and 2.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator or sub-investigator, the participant is capable of understanding and complying with protocol requirements.
2. The participant signs and dates a written, informed consent form prior to the initiation of any study procedures.
3. The participant is a healthy Japanese adult male, aged 20 to 60 years, inclusive, at the time of informed consent.
4. The participant weighs at least 50 kilogram (kg) and has a body mass index (BMI) from 18.5 to 25.0 kilogram per square meter (kg/m^2), inclusive at Screening.
5. The participant must be a current nonsmoker who has not used tobacco- or nicotine-containing products (example, nicotine patch) for at least 6 months prior to the start of study drug administration in Period 1.
6. The participant must be judged to be in good health by the investigator, based on clinical evaluations including laboratory safety tests, medical history, physical examination, 12-lead electrocardiogram (ECG), and vital sign measurements performed at the Screening Visit and prior to the start of study drug administration in Period 1.

Exclusion Criteria:

1. The participant has received any investigational compound within 16 weeks (112 days) prior to the start of study drug administration in Period 1.
2. The participant has received TAK-438 in a previous clinical study or as a therapeutic agent.
3. The participant is an immediate family member of or a study site employee, or is in a dependent relationship with a study site employee who is involved in the conduct of this study (example, spouse, parent, child, sibling) or may consent under duress.
4. The participant has uncontrolled, clinically significant neurologic, cardiovascular, pulmonary, hepatic, renal, metabolic, gastrointestinal, urologic, or endocrine disease or other abnormality (other than the disease being studied), which may impact the ability of the participant to participate in the study or potentially confound its results.
5. The participant has hypersensitivity to any component of TAK-438 OD tablet or TAK-438 tablet.
6. The participant has a positive urine drug result for drugs of abuse at Screening.
7. The participant has a history of drug or alcohol abuse within 2 years prior to the Screening visit or is unwilling to agree to abstain from alcohol and drugs throughout the study.
8. The participant has taken any excluded medication, supplements, or food products during the specified time periods.
9. The participant has current or recent (within 6 months) gastrointestinal disease that would be expected to influence the absorption of drugs (ie, a history of malabsorption, esophageal reflux, peptic ulcer disease, erosive esophagitis), frequent (more than once per week) occurrence of heartburn, or any surgical intervention.
10. The participant has a history of cancer, except basal cell carcinoma which has been in remission for at least 5 years prior to Day 1.
11. The participant has a positive test result for hepatitis B virus surface antigen (HBsAg), hepatitis C virus (HCV) antibody, human immunodeficiency virus (HIV) antibody/antigen, or serological reactions for syphilis at Screening.
12. The participant has poor peripheral venous access.
13. The participant has undergone whole blood collection of at least 200 milliliter (mL) within 4 weeks (28 days) or at least 400 mL within 12 weeks (84 days) prior to the start of study drug administration in Period 1.
14. The participant has undergone whole blood collection of at least 800 mL in total within 52 weeks (364 days) prior to the start of study drug administration in Period 1.
15. The participant has undergone blood component collection within 2 weeks (14 days) prior to the start of study drug administration in Period 1.
16. The participant has a Screening or Check-in (Day -1) ECG that was abnormal (clinically significant).
17. The participant has abnormal Screening laboratory values that suggest a clinically significant underlying disease or participant with the following laboratory abnormalities: alanine aminotransferase (ALT) or aspartate aminotransferase (AST) above the upper limits of normal (ULN).
18. The participant who, in the opinion of the investigator or sub-investigator, is unlikely to comply with the protocol or is unsuitable for any other reason.

Ages: 20 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 48 (Actual)
Dates: Start 2019-01-30 (Actual); Primary Completion 2019-03-12 (Actual); Study Completion 2019-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Sekino Clinical Pharmacology Clininc, Toshima-ku, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in Japan from 30 January 2019 to 12 March 2019.
Pre-assignment Details: Healthy Japanese male participants were enrolled in 1 of the 2 treatment sequences to receive TAK-438 OD 20 milligram (mg) or TAK-438 20 mg with or without water in Study 1, and TAK-438 OD 20 mg or TAK-438 20 mg with water in Study 2. Study was completed with Pilot study since results from interim analysis satisfied the criteria of bioequivalence.
Groups:
- Pilot BE Study 1, Sequence A: TAK-438 OD 20 mg + TAK-438 20 mg: TAK-438 orally disintegrating (OD) 20 mg, tablet, orally without water under fasted condition, once on Day 1 of Period 1, followed by a washout period of at least 7 days, further followed by TAK-438 20 mg, tablet, orally with water under fasted condition, once on Day 1 of Period 2.
- Pilot BE Study 1, Sequence B: TAK-438 20 mg + TAK-438 OD 20 mg: TAK-438 20 mg, tablet, orally with water under fasted condition, once on Day 1 of Period 1 followed by a washout period of at least 7 days, further followed TAK-438 OD 20 mg, tablet, orally without water under fasted condition, once on Day 1 of Period 2.
- Pilot BE Study 2, Sequence C: TAK-438 OD 20 mg + TAK-438 20 mg: TAK-438 OD 20 mg, tablet, orally with water under fasted condition, once on Day 1 of Period 1, followed by a washout period of at least 7 days, further followed by TAK-438 20 mg tablet, orally with water under fasted condition, once on Day 1 of Period 2.
- Pilot BE Study 2, Sequence D: TAK-438 20 mg + TAK-438 OD 20 mg: TAK-438 20 mg, tablet, orally with water under fasted condition, once on Day 1 of Period 1, followed by a washout period of at least 7 days, further followed by TAK-438 OD 20 mg tablet, orally with water under fasted condition, once on Day 1 of Period 2.
Period: Overall Study
Arm/Group | Pilot BE Study 1, Sequence A: TAK-438 OD 20 mg + TAK-438 20 mg | Pilot BE Study 1, Sequence B: TAK-438 20 mg + TAK-438 OD 20 mg | Pilot BE Study 2, Sequence C: TAK-438 OD 20 mg + TAK-438 20 mg | Pilot BE Study 2, Sequence D: TAK-438 20 mg + TAK-438 OD 20 mg
Started | 12 | 12 | 12 | 12
Completed (Here, completed means completion of all periods, that means Period 1, Washout period, and Period 2.) | 12 | 12 | 12 | 12
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set was defined as all participants who received at least one dose of study drug.
Groups:
- Pilot BE Study 1, Sequence A: TAK-438 OD 20 mg + TAK-438 20 mg: TAK-438 OD 20 mg, tablet, orally without water under fasted condition, once on Day 1 of Period 1, followed by a washout period of at least 7 days, further followed by TAK-438 20 mg, tablet, orally with water under fasted condition, once on Day 1 of Period 2.
- Total: Total of all reporting groups
Arm/Group | Pilot BE Study 1, Sequence A: TAK-438 OD 20 mg + TAK-438 20 mg | Pilot BE Study 1, Sequence B: TAK-438 20 mg + TAK-438 OD 20 mg | Pilot BE Study 2, Sequence C: TAK-438 OD 20 mg + TAK-438 20 mg | Pilot BE Study 2, Sequence D: TAK-438 20 mg + TAK-438 OD 20 mg | Total
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.1 (3.87) | 26.0 (6.74) | 26.5 (7.19) | 26.0 (6.76) | 25.1 (6.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 12 | 12 | 12 | 12 | 48
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 12 | 12 | 12 | 12 | 48
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 171.8 (4.00) | 170.0 (6.52) | 173.9 (4.32) | 172.2 (6.94) | 172.0 (5.59)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 59.83 (4.672) | 60.95 (4.720) | 63.29 (4.860) | 65.44 (6.716) | 62.38 (5.586)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 20.28 (1.817) | 21.15 (1.829) | 20.94 (1.781) | 22.03 (1.043) | 21.10 (1.718)
Caffeine Consumption [Count of Participants; unit: Participants]
  Had caffeine consumption | 2 | 1 | 4 | 4 | 11
  Had no caffeine consumption | 10 | 11 | 8 | 8 | 37
Alcohol Consumption [Count of Participants; unit: Participants]
  Drank a few times per week | 0 | 2 | 0 | 1 | 3
  Drank a few times per month | 6 | 3 | 4 | 1 | 14
  Never drank | 6 | 7 | 8 | 10 | 31
Smoking Classification [Count of Participants; unit: Participants]
  Never smoked | 11 | 11 | 10 | 11 | 43
  Former smoker | 1 | 1 | 2 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: AUClast: Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Plasma Concentration for TAK-438 Free Base (TAK-438F)
Time Frame: Day 1 pre-dose and at multiple time points (up to 48 hours; 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36 and 48 hours) post-dose
Population: The pharmacokinetic (PK) analysis set was defined as all participants who received at least one dose of study drug, and whose PK data were evaluable.
Measure: Geometric Mean (Standard Deviation); unit: hour*nanogram per milliliter (h*ng/mL)
Groups:
- Pilot BE Study 1: TAK-438 OD 20 mg: TAK-438 OD 20 mg, tablet, orally without water under fasted condition, once on Day 1 of either Period 1 or 2.
- Pilot BE Study 1: TAK-438 20 mg; Pilot BE Study 2: TAK-438 20 mg: TAK-438 20 mg, tablet, orally with water under fasted condition, once on Day 1 of either Period 1 or 2.
- Pilot BE Study 2: TAK-438 OD 20 mg: TAK-438 OD 20 mg, tablet, orally with water under fasted condition, once on Day 1 of either Period 1 or 2.
Arm/Group | Pilot BE Study 1: TAK-438 OD 20 mg | Pilot BE Study 1: TAK-438 20 mg | Pilot BE Study 2: TAK-438 OD 20 mg | Pilot BE Study 2: TAK-438 20 mg
Number analyzed (Participants) | 24 | 24 | 24 | 24
hour*nanogram per milliliter (h*ng/mL) | 190.2 (67.984) | 194.3 (67.693) | 201.6 (81.799) | 201.2 (75.813)
Statistical Analysis 1: Comparison: Pilot BE Study 1: TAK-438 OD 20 mg vs Pilot BE Study 1: TAK-438 20 mg; Test type: Equivalence — For log-transformed (natural log) AUClast, the two-sided 90% CI of the difference in the least square means (LS-Means) between the formulations (TAK-438 OD tablet-TAK-438 tablet) was provided using the ANOVA model; LS-Means Difference = -0.0211, 90% CI 2-sided [-0.0752 to 0.0329]
Statistical Analysis 2: Comparison: Pilot BE Study 2: TAK-438 OD 20 mg vs Pilot BE Study 2: TAK-438 20 mg; Test type: Equivalence — For log-transformed (natural log) AUClast, the two-sided 90% CI of the difference in the LS-Means between the formulations (TAK-438 OD tablet-TAK-438 tablet) was provided using the ANOVA model; LS-Means Difference = 0.0019, 90% CI 2-sided [-0.0778 to 0.0815]

2. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for TAK-438F
Time Frame: as for outcome 1
Population: The PK analysis set was defined as all participants who received at least one dose of study drug, and whose PK data were evaluable.
Measure: Geometric Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Pilot BE Study 1: TAK-438 OD 20 mg | Pilot BE Study 1: TAK-438 20 mg | Pilot BE Study 2: TAK-438 OD 20 mg | Pilot BE Study 2: TAK-438 20 mg
Number analyzed (Participants) | 24 | 24 | 24 | 24
nanogram per milliliter (ng/mL) | 22.62 (7.8152) | 24.26 (8.0676) | 21.85 (7.7286) | 23.70 (8.5998)
Statistical Analysis 1: Comparison: Pilot BE Study 1: TAK-438 OD 20 mg vs Pilot BE Study 1: TAK-438 20 mg; Test type: Equivalence — For log-transformed (natural log) Cmax, the two-sided 90% CI of the difference in the LS-Means between the formulations (TAK-438 OD tablet-TAK-438 tablet) was provided using the ANOVA model; LS-Means Difference = -0.0698, 90% CI 2-sided [-0.1404 to 0.0008]
Statistical Analysis 2: Comparison: Pilot BE Study 2: TAK-438 OD 20 mg vs Pilot BE Study 2: TAK-438 20 mg; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; LS-Means Difference = -0.0811, 90% CI 2-sided [-0.1658 to 0.0036]

3. Secondary Outcome: AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for TAK-438F
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Pilot BE Study 1: TAK-438 OD 20 mg | Pilot BE Study 1: TAK-438 20 mg | Pilot BE Study 2: TAK-438 OD 20 mg | Pilot BE Study 2: TAK-438 20 mg
Number analyzed (Participants) | 24 | 24 | 24 | 24
h*ng/mL | 192.5 (68.755) | 196.4 (68.436) | 204.3 (83.014) | 203.6 (77.630)
Statistical Analysis 1: Comparison: Pilot BE Study 1: TAK-438 OD 20 mg vs Pilot BE Study 1: TAK-438 20 mg; Test type: Equivalence — For log-transformed (natural log) AUC∞, the two-sided 90% CI of the difference in the LS-Means between the formulations (TAK-438 OD tablet-TAK-438 tablet) was provided using the ANOVA model; LS-Means Difference = -0.0199, 90% CI 2-sided [-0.0731 to 0.0333]
Statistical Analysis 2: Comparison: Pilot BE Study 2: TAK-438 OD 20 mg vs Pilot BE Study 2: TAK-438 20 mg; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; LS-Means Difference = 0.0035, 90% CI 2-sided [-0.0760 to 0.0830]

4. Secondary Outcome: Tmax: Time of First Occurrence of Maximum Plasma Concentration (Cmax) for TAK-438F
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Full Range); unit: hour
Arm/Group | Pilot BE Study 1: TAK-438 OD 20 mg | Pilot BE Study 1: TAK-438 20 mg | Pilot BE Study 2: TAK-438 OD 20 mg | Pilot BE Study 2: TAK-438 20 mg
Number analyzed (Participants) | 24 | 24 | 24 | 24
hour | 2.000 [1.00 to 4.00] | 1.750 [1.00 to 3.00] | 2.000 [1.00 to 4.00] | 2.000 [1.00 to 4.00]
Statistical Analysis 1: Comparison: Pilot BE Study 1: TAK-438 OD 20 mg vs Pilot BE Study 1: TAK-438 20 mg; Test type: Equivalence — For log-transformed (natural log) Tmax, the two-sided 90% CI of the difference in the LS-Means between the formulations (TAK-438 OD tablet-TAK-438 tablet) was provided using the ANOVA model; LS-Means Difference = 0.1902, 90% CI 2-sided [0.0199 to 0.3605]
Statistical Analysis 2: Comparison: Pilot BE Study 2: TAK-438 OD 20 mg vs Pilot BE Study 2: TAK-438 20 mg; Test type: Equivalence — [test comment as in outcome 4, analysis 1]; LS-Means Difference = 0.2142, 90% CI 2-sided [0.0558 to 0.3725]

5. Secondary Outcome: MRT∞,ev: Mean Residence Time After Extravascular Administration From Time 0 to Infinity for TAK-438F
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Pilot BE Study 1: TAK-438 OD 20 mg | Pilot BE Study 1: TAK-438 20 mg | Pilot BE Study 2: TAK-438 OD 20 mg | Pilot BE Study 2: TAK-438 20 mg
Number analyzed (Participants) | 24 | 24 | 24 | 24
hour | 9.576 (1.1807) | 9.258 (0.91125) | 9.831 (1.3506) | 9.544 (1.4121)
Statistical Analysis 1: Comparison: Pilot BE Study 1: TAK-438 OD 20 mg vs Pilot BE Study 1: TAK-438 20 mg; Test type: Equivalence — For log-transformed (natural log) MRT∞,ev, the two-sided 90% CI of the difference in the LS-Means between the formulations (TAK-438 OD tablet-TAK-438 tablet) was provided using the ANOVA model; LS-Means Difference = 0.0311, 90% CI 2-sided [0.0022 to 0.0599]
Statistical Analysis 2: Comparison: Pilot BE Study 2: TAK-438 OD 20 mg vs Pilot BE Study 2: TAK-438 20 mg; Test type: Equivalence — [test comment as in outcome 5, analysis 1]; LS-Means Difference = 0.0306, 90% CI 2-sided [-0.0003 to 0.0616]

6. Secondary Outcome: λz: Terminal Disposition Phase Rate Constant for TAK-438F
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: per hour (1/hour)
Arm/Group | Pilot BE Study 1: TAK-438 OD 20 mg | Pilot BE Study 1: TAK-438 20 mg | Pilot BE Study 2: TAK-438 OD 20 mg | Pilot BE Study 2: TAK-438 20 mg
Number analyzed (Participants) | 24 | 24 | 24 | 24
per hour (1/hour) | 0.1014 (0.014441) | 0.09903 (0.011269) | 0.09807 (0.013021) | 0.09989 (0.016690)
Statistical Analysis 1: Comparison: Pilot BE Study 1: TAK-438 OD 20 mg vs Pilot BE Study 1: TAK-438 20 mg; Test type: Equivalence — For log-transformed (natural log) λz, the two-sided 90% CI of the difference in the LS-Means between the formulations (TAK-438 OD tablet-TAK-438 tablet) was provided using the ANOVA model; LS-Means Difference = 0.0209, 90% CI 2-sided [-0.0112 to 0.0530]
Statistical Analysis 2: Comparison: Pilot BE Study 2: TAK-438 OD 20 mg vs Pilot BE Study 2: TAK-438 20 mg; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; LS-Means Difference = -0.0135, 90% CI 2-sided [-0.0508 to 0.0238]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) are adverse events (AE) that started after the first dose of study drug until Day 3 in Period 2 (up to Day 13)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Pilot BE Study 1: TAK-438 OD 20 mg | Pilot BE Study 1: TAK-438 20 mg | Pilot BE Study 2: TAK-438 OD 20 mg | Pilot BE Study 2: TAK-438 20 mg
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Study Protocol (2018-12-12): https://cdn.clinicaltrials.gov/large-docs/93/NCT03808493/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-27): https://cdn.clinicaltrials.gov/large-docs/93/NCT03808493/SAP_001.pdf